CLINICAL TRIAL: NCT05257148
Title: Open-label, Multicenter, Multinational, Interventional Clinical Trial to Assess Effectiveness and SAfety of the Extemporaneous Combination of Nebivolol and Zofenopril Calcium in Grade 1 to 2 Hypertensive patIents Versus Each mOnotherapy
Brief Title: Effectiveness and Safety of Combination of Nebivolol and Zofenopril in Hypertensive patIents Versus Each Monotherapy
Acronym: Masaccio
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEIN/19/ZoNe-HYP/001; 2020-002340-23 (EudraCT Number)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-11

CONDITIONS: Hypertension
Keywords: Hypertension; Combination Therapy; Zofenopril; Nebivolol; Fixed Dose Combination
MeSH Terms: conditions — Hypertension | interventions — zofenopril; Nebivolol

STUDY DESIGN:
Intervention Model Description: Open Label, two period study. Patients eligible from screening will enter the run-in period on the same day. Patients previously receiving Zofenopril or any other ACE-inhibitor will enter into the run-in period with Zofenopril monotherapy while patients receiving Nebivolol or any other Beta Blockers will enter into the Run-in period with Nebivolol monotherapy in a 1:1 ratio.
  Only patients with uncontrolled BP (sitting Systolic Blood Pressure/Diastolic Blood Pressure>130/80 mmHg) and whose adherence to the treatment ranges from 80% to 120%, will enter the assessment period to receive the extemporaneous combination of NEB and ZOF; while the patients with controlled sitting BP (Systolic Blood Pressure/Diastolic Blood Pressure ≤130/80 mmHg) and/or the patients who do not tolerate the treatment and patients with uncontrolled BP whose adherence to the therapy do not range from 80% to 120%, will be withdrawn from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zofenopril arm (Active Comparator): MONOTHERAPY PERIOD (one month): patients will be treated with Zofenopril 30 mg. COMBINATION THERAPY PERIOD (two months) patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Nebivolol 5mg
  Interventions: Drug: Zofenopril 30 mg; Drug: Zofenopril 30 mg + Nebivolol 5 mg
- Nebivolol arm (Active Comparator): MONOTHERAPY PERIOD (one month): patients will be treated with Nebivolol 5 mg. COMBINATION THERAPY PERIOD (two months) patients will be treated with the extemporaneous combination of Zofenopril 30 mg and Nebivolol 5 mg
  Interventions: Drug: Nebivolol 5 mg; Drug: Zofenopril 30 mg + Nebivolol 5 mg

INTERVENTIONS:
Drug: Zofenopril 30 mg — Film-Coated tablets administered as one single dose to be taken in the morning (from 6 am to 10 am) with no restriction on food intake
  Arms: Zofenopril arm
Drug: Nebivolol 5 mg — Tablet administered as one single dose to be taken in the morning (from 6 am to 10 am) with no restriction on food intake
  Arms: Nebivolol arm
Drug: Zofenopril 30 mg + Nebivolol 5 mg — Both Film coated tablets of Zofenopril 30 mg and Nebivolol 5 mg Tablets will be taken in the morning (from 6 am to 10 am) with no restriction on food intake

SUMMARY:
Open-label, interventional clinical trial to assess effectiveness and safety of the extemporaneous combination of nebivolol and zofenopril calcium in grade 1 to 2 hypertensive patients versus each monotherapy

DETAILED DESCRIPTION:
This is a study with 2 periods (a run-in period of 4 weeks and an assessment period of 8 weeks). Grade 1-2 hypertensive patients (blood pressure [BP] ranging from ≥140/90 mmHg to ≤179/109 mmHg) on treatment with any angiotensin converting enzyme-inhibitors (ACEi) or beta blockers (BBs) including ZOF 30 mg or NEB 5 mg respectively will be screened for eligibility (Visit 1).

On the same day, the eligible patients will enter into a run-in period after Screening, during which:

* Patients on ZOF 30 mg or NEB 5 mg will continue the same therapy for 4 weeks
* Patients on any other ACE-i will be assigned to monotherapy with ZOF 30 mg while patients on any other BB will be assigned to monotherapy with NEB 5 mg, respectively, for 4 weeks.

After the 4 weeks of monotherapy in the run-in period, if BP at Visit 2, remains uncontrolled (sitting Systolic Blood Pressure/Diastolic Blood Pressure >130/80 mmHg) despite an adherence to the treatments ranging from 80% to 120%, the patients will start treatment (Week 0, Visit 2) with the extemporaneous combination of NEB 5 mg/ZOF 30 mg (NEB/ZOF) and will be assessed for further 8 weeks (assessment period).

If the patients, at Visit 2 after the Run-In period, have controlled BP (sitting Systolic Blood Pressure/Diastolic Blood Pressure ≤130/80 mmHg), and/or do not tolerate the treatment, and/or do not maintain the adherence to the therapy (range from 80% to 120%), these patients will not be continued further in the study.

At the end of the assessment period (Visit 3) the anti-hypertensive effect of the extemporaneous combination of NEB 5 mg and ZOF 30 mg will be evaluated.

A total number of 290 patients will be screened considering 25% of drop-out rate, to obtain approximately 216 completed patients at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Caucasian uncontrolled hypertensive patients (see definition in criterion 3) ≥18 and <65 years of age, in monotherapy either with ACE-i or BBs since at least 1 month, at Screening (Visit 1)
2. Patients are able to understand and have freely given written informed consent at Screening
3. Patients with mean sitting Systolic Blood Pressure ≥140 mmHg and ≤179 mmHg and/or mean sitting Diastolic Blood Pressure ≥ 90 mmHg and ≤109 mmHg at Screening (Visit 1)
4. Patient who are able to comply with all study procedures and who are available for the duration of the study
5. Ability to take oral medication and willing to adhere to the drug regimen
6. A female patient of childbearing potential is eligible to participate if she is not pregnant, or not breastfeeding. A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile. Women of childbearing potential must agree to use of highly effective contraception (eg, method of birth control throughout the study period and for 4 weeks after study completion defined as a method which results in a failure rate of less than 1% per year) and also must refrain from donating or storing eggs during this time. Highly effective contraception methods can be: a Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) b Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) c Intrauterine device (IUD) d Intrauterine hormone-releasing system (IUS) e Bilateral tubal occlusion f Vasectomized partner (provided that partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success)
7. A male patient with female partner must agree to use contraception during the whole study period and for at least 1 week after the last dose of study treatment and refrain from donating sperms during this period.

Exclusion Criteria:

1. Known contraindications, allergies, or hypersensitivities to any of the study medications or excipient as outlined in the investigators brochures (IBs), summary of product characteristics (SmPCs) or local package inserts for NEB and ZOF
2. Patients with serious disorders (in the opinion of the Investigator) which may limit the ability to evaluate the efficacy or safety of the tested medications, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine/ or metabolic, hematological, or oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic patients
3. Patients having a history of the following within the last 6 months:

   myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, bypass surgery, heart failure, hypertensive encephalopathy, cerebrovascular accident (stroke), or transient ischemic attack
4. Patients with secondary hypertension of any etiology such as renal diseases, pheochromocytoma, or Cushing's syndrome
5. Patients with severe heart failure (New York Heart Association classification III-IV), a narrowing of the aortic or bicuspid valve, an obstruction of cardiac outflow (obstructive, hypertrophic cardiomyopathy) or symptomatic coronary disease
6. Patients with clinical evidence of renal disease as per the Investigator's judgement (including renovascular occlusive disease, nephrectomy and/or renal transplant, bilateral renal artery stenosis or unilateral renal artery stenosis in a solitary kidney, or severe renal impairment)
7. History of angioneurotic edema
8. Patients with clinically relevant hepatic impairment
9. Patients with sick sinus syndrome, including sino-atrial block
10. Patients with second- or third-degree heart block (without a pacemaker)
11. History of bronchospasm and bronchial asthma
12. Patients with bradycardia (heart rate <60 bpm)
13. Patient with metabolic acidosis
14. Patients with severe peripheral circulatory disturbances
15. Participation in another study within the last 4 weeks
16. Patients with diseases that, in the opinion of the Investigator, prevent a careful adherence to the protocol
17. Pregnant and breastfeeding women. A pregnancy test will be performed on all women of childbearing potential at each study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Volpe, Professor, Principal Investigator — University "Sapienza" Rome
Locations (1):
- Istituto Clinico Humanitas, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started on 26 May 2021 and terminated on 22 December 2021 296 patients were screened for the study. 283 patients entered the run-in period and were assigned for monotherapy to Nebivolol (NEB) 5 mg or Zofenopril (ZOF) 30 mg. Of the 269 completed patients in monotherapy, 246 were assigned to combination therapy and 238 competed the study
Pre-assignment Details: Run-in period (Week -4 to Week 0):
  • Patients on ZOF 30 mg or NEB 5 mg continued the same therapy. Patients on any other angiotensin I-converting enzyme (ACE-i) were assigned to monotherapy with ZOF 30 mg and the patients on any other betablocker (BB) were assigned to monotherapy with NEB 5 mg, respectively.
Period: Run in
Arm/Group | Zofenopril Arm | Nebivolol Arm
Started | 137 | 146
Completed | 130 | 139
Not Completed | 7 | 7
Period: Assessment
Arm/Group | Zofenopril Arm | Nebivolol Arm
Started | 119 (Number of subjects starting this period is not consistent with the number completing the preceding period because after Run-in Period, Patients with controlled BP [sitting Systolic Blood Pressure (SBP / DBP ≤ 130/80 mmHg)] at Week 0 (Visit 2), patients with uncontrolled BP (sitting SBP / DBP > 130/80 mmHg) whose adherence to the treatment was not included from 80% to 120%, or patients who could not tolerate mono therapies, were discontinued from the study and excluded from the Assessment Period.) | 127 (The number of subjects starting this period is not consistent with the number completing the preceding period because after Run-in Period, Patients with controlled BP (sitting SBP / DBP ≤ 130/80 mmHg) at Week 0 (Visit 2), patients with uncontrolled BP (sitting SBP / DBP > 130/80 mmHg) whose adherence to the treatment was not included from 80% to 120%, or patients who could not tolerate one of the mono therapies were discontinued from the study and excluded from the Assessment Period.)
Completed | 115 | 123
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Intentio to treat population
Groups:
- COMBINATION THERAPY PERIOD Zofenopril 30mg/Nebivolol 5mg: During the assessment period of 8 weeks, the eligible patients (uncontrolled hypertension with sitting BP of SBP/DBP > 130/80 mmHg, who tolerated the treatment and whose adherence to the therapies ranged from 80% to 120%) received a combination of NEB 5 mg and ZOF 30 mg to be taken orally once daily.
Arm/Group | COMBINATION THERAPY PERIOD Zofenopril 30mg/Nebivolol 5mg
Number analyzed (Participants) | 246
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 246
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 246
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 16
  Poland | 230

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting DBP Between Week 0 (Visit 2) and Week 8 (Visit 3)
Description: To assess the antihypertensive efficacy of the extemporaneous combination of Nebivolol (NEB) 5 mg and Zofenopril (ZOF) 30 mg in lowering sitting diastolic blood pressure (DBP) from baseline (Visit 2) after 8 weeks of treatment (Visit 3), in patients with uncontrolled blood pressure (BP) who were previously treated with NEB or ZOF monotherapies for at least 4 weeks.
Time Frame: From Baseline (Week 0 - Visit 2) to week 8 (Visit 3)
Population: Intention to Treat Population composed by all patients who were enrolled and received at least 1 dose of the combination therapy and have at least 1 post baseline safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | COMBINATION THERAPY PERIOD Zofenopril 30mg/Nebivolol 5mg
Number analyzed (Participants) | 241
mmHg | -9.3 (8.94)
Statistical Analysis 1: Comparison: COMBINATION THERAPY PERIOD Zofenopril 30mg/Nebivolol 5mg; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -9.3

ADVERSE EVENTS:
Time Frame: From Informed Consent signature at screening visit (Visit 1) occurring 4 week previous than Baseline assessment (Week 0 - Visit 2) to last visit at Week 8 (Visit 3) for an average of 12 weeks. Furthermore patients having any ongoing Adverse Event/Serious Adverse Event at the end of the treatment (Week 8 - Visit 3), will be followed for further 2 weeks via a phone call to check about the status of the Adverse Events/Serious Adverse Events, extending the time frame to a total of 14 weeks.
Groups:
- Zofenopril 30mg MONOTHERAPYPERIOD: Adverse events occurred to Enrolled population that received Zofenopril 30mg during the Run-in period of 4 Weeks, from Screening visit (Visit 1 - Week -4) to Visit 2 (Week 0).
- Nebivolol 5mg MONOTHERAPYPERIOD: Adverse events occurred to Enrolled population that received Nebivolol 5mg during the Run-in period of 4 Weeks, from Screening visit (Visit 1 - Week -4) to Visit 2 (Week 0).
- Zofenopril 30mg/Nebivolol 5mg COMBINATION THERAPY PERIOD: Adverse events occurred to Enrolled population that received combination therapy during the assessment period of 8 weeks from Visit 2 (Week 0) to visit 3 (Week 8).
Arm/Group | Zofenopril 30mg MONOTHERAPYPERIOD | Nebivolol 5mg MONOTHERAPYPERIOD | Zofenopril 30mg/Nebivolol 5mg COMBINATION THERAPY PERIOD
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/146 | 0/246
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/146 | 0/246
Other Adverse Events (participants affected / at risk) | 9/137 | 2/146 | 18/246
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zofenopril 30mg MONOTHERAPYPERIOD (N=137) | Nebivolol 5mg MONOTHERAPYPERIOD (N=146) | Zofenopril 30mg/Nebivolol 5mg COMBINATION THERAPY PERIOD (N=246)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 — Worsening
hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 — Worsening
Mixed Hyperlipidemia (Metabolism and nutrition disorders) | 2 | 0 (0) | 1 — Acquired
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 — Worsening
Headache (Nervous system disorders) | 1 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose Tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infections (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Cardiac Discomfort (Cardiac disorders) | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT05257148/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05257148/SAP_001.pdf